CLINICAL TRIAL: NCT00964301
Title: Telemedicine Education for Rural Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110807
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Asthma; Low-income; Quality of life; Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Participants, caregivers and school nurse will attend telemedicine education sessions at school.
  Interventions: Other: Telemedicine Education
- Usual care (Active Comparator): Usual care participant will receive routine care from their primary care provider.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Telemedicine Education — Student Asthma Education. Each student will engage in 6 age-appropriate sessions on various aspects of asthma health.
  Caregiver Asthma Education. The primary caregiver will engage in 2 asthma education sessions.
  School Nurse Asthma Education. School nurses will participate in 2 sessions.
  Primary Care Provider (PCP) Communication. The PCP of the intervention group participant will be notified of his/her patient's baseline asthma assessment. They will receive updates summarizing each telemedicine intervention.
  Arms: Intervention Group
Other: Usual care — Participants will receive asthma care by their PCP with no education sessions or PCP communications by the research staff.
  Arms: Usual care

SUMMARY:
The investigators will implement an interactive school-based telemedicine education program for rural low-income, minority children with asthma, their caregivers, and school nurses in the Delta region of Arkansas.

Specific aims:

1. The investigators will examine changes in asthma symptoms control and other health outcomes such as activity levels and family/child emotional health in the intervention group compared to a usual care group.
2. The investigators will examine changes in asthma knowledge, self-efficacy, and quality of life in the intervention participants and their caregivers compared to a usual care group.

DETAILED DESCRIPTION:
The investigators will conduct a prospective study to examine the impact of an interactive, telemedicine asthma intervention among children living in the rural Delta region of Arkansas.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be English-speaking children ages 7-17 years with physician-diagnosed asthma and/or active symptoms in the previous 12 months.
* Active symptoms include one or more of the following:

  * experience daytime wheezing, shortness of breath, and/or coughing two or more times a week for the last 4 weeks;
  * nighttime wheezing, shortness of breath and/or cough more than once a week;
  * take asthma medication more than two days a week;
  * have been treated in a hospital or emergency department two or more times in the last two years for asthma symptoms;
  * have been treated in a hospital or emergency department two or more times in the last two years for asthma symptoms have episodes of asthma-like symptoms when playing/exercising.
* Potentially eligible participants will be screened using an asthma screener to confirm eligibility.

Exclusion Criteria:

* Children with significant underlying respiratory disease other than asthma (such as cystic fibrosis) or significant co-morbid conditions (such as severe developmental delay or cerebral palsy) will be excluded from the study.
* The primary caregiver and child will be asked questions via telephone interview about how asthma affects the child every day. Children with no telephone number or contact telephone number will be excluded.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The investigators will examine changes in asthma symptoms control and health outcomes in the intervention group compared to a usual care group. | One year

SECONDARY OUTCOMES:
The investigators will examine changes in asthma knowledge, self-efficacy, and quality of life of the intervention participants and their caregivers compared to a usual care group. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, M.D., FAAP, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Perry TT, Vargas PA, McCracken A, Jones SM. Underdiagnosed and uncontrolled asthma: findings in rural schoolchildren from the Delta region of Arkansas. Ann Allergy Asthma Immunol. 2008 Oct;101(4):375-81. doi: 10.1016/S1081-1206(10)60313-4. PMID 18939725
- [Background] Perry TT, Vargas PA, Brown RH et al. Asthma morbidity in high risk rural children in the delta region of Arkansas. J Allergy Clin Immunol. 2008;121:S231
- [Background] Dey AN, Schiller JS, Tai DA. Summary health statistics for U.S. children: National Health Interview Survey, 2002. Vital Health Stat 10. 2004 Mar;(221):1-78. PMID 15791897
- [Background] Weitzman M, Gortmaker S, Sobol A. Racial, social, and environmental risks for childhood asthma. Am J Dis Child. 1990 Nov;144(11):1189-94. doi: 10.1001/archpedi.1990.02150350021016. PMID 2239856
- [Background] Yeatts K, Davis KJ, Sotir M, Herget C, Shy C. Who gets diagnosed with asthma? Frequent wheeze among adolescents with and without a diagnosis of asthma. Pediatrics. 2003 May;111(5 Pt 1):1046-54. doi: 10.1542/peds.111.5.1046. PMID 12728087
- [Background] Chrischilles E, Ahrens R, Kuehl A, Kelly K, Thorne P, Burmeister L, Merchant J. Asthma prevalence and morbidity among rural Iowa schoolchildren. J Allergy Clin Immunol. 2004 Jan;113(1):66-71. doi: 10.1016/j.jaci.2003.09.037. PMID 14713909
- [Background] Vargas PA, Simpson PM, Gary Wheeler J, Goel R, Feild CR, Tilford JM, Jones SM. Characteristics of children with asthma who are enrolled in a Head Start program. J Allergy Clin Immunol. 2004 Sep;114(3):499-504. doi: 10.1016/j.jaci.2004.05.025. PMID 15356547
- [Background] Vargas PA, Simpson PM, Bushmiaer M, Goel R, Jones CA, Magee JS, Feild CR, Jones SM. Symptom profile and asthma control in school-aged children. Ann Allergy Asthma Immunol. 2006 Jun;96(6):787-93. doi: 10.1016/S1081-1206(10)61340-3. PMID 16802765
- [Background] Nash C, Ochoa ER. Arkansas Racial and Ethnic Health Disparity Study Report. Little Rock, AR: Arkansas Minority Health Commission, 2004.
- [Background] National Asthma Education and Prevention Program Expert Panel Report 3: Guidelines for the Diagnosis and Management of Asthma. National Heart Lung and Blood Insitutute. 2007.
- [Background] Butz A, Pham L, Lewis L, Lewis C, Hill K, Walker J, Winkelstein M. Rural children with asthma: impact of a parent and child asthma education program. J Asthma. 2005 Dec;42(10):813-21. doi: 10.1080/02770900500369850. PMID 16393717
- [Background] Bursch B, Schwankovsky L, Gilbert J, Zeiger R. Construction and validation of four childhood asthma self-management scales: parent barriers, child and parent self-efficacy, and parent belief in treatment efficacy. J Asthma. 1999;36(1):115-28. doi: 10.3109/02770909909065155. PMID 10077141